CLINICAL TRIAL: NCT03582306
Title: Exploring the Effects of a High Chlorophyll Dietary Intervention to Reduce Colon Cancer Risk in Adults: The Meat and Three Greens Feasibility Trial
Brief Title: Exploring the Effects of a High Chlorophyll Dietary Intervention to Reduce Colon Cancer Risk in Adults
Acronym: M3G
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Andrew Fruge, Assistant Professor and Director, Didactic Program in Dietetics, Auburn University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AU-18-208
Record Dates: First submitted 2018-06-10; First posted 2018-07-11 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Colon Cancer Prevention
Keywords: colon cancer; dietary intervention; vegetables; microbiota
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: 4 week intervention and control periods will be delivered and separated by a 4 week washout. The order of intervention and control periods will be randomly allocated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High chlorophyll diet - intervention 1st (Experimental): Participants will complete the 4 week intervention, 4 week washout, then 4 week control period (monitor only)
  Interventions: Behavioral: High chlorophyll diet - intervention 1st
- High chlorophyll diet - control 1st (Experimental): Participants will complete the 4 week control period (monitor only), 4 week washout, then 4 week intervention
  Interventions: Behavioral: High chlorophyll diet - control 1st

INTERVENTIONS:
Behavioral: High chlorophyll diet - intervention 1st — Participants will be provided frozen dark leafy green vegetables, and counseled to consume 1 cup cooked dark green leafy vegetables (2 servings) daily over the 4 week period while maintaining their normal red meat intake. This will occur during the first 4 week period of the study.
  Other Names: High green leafy vegetable diet
  Arms: High chlorophyll diet - intervention 1st
Behavioral: High chlorophyll diet - control 1st — Participants will be provided frozen dark leafy green vegetables, and counseled to consume 1 cup cooked dark green leafy vegetables (2 servings) daily over the 4 week period while maintaining their normal red meat intake. This will occur during the last 4 week period of the study.
  Other Names: High green leafy vegetable diet
  Arms: High chlorophyll diet - control 1st

SUMMARY:
Colon cancer is the third most common cancer in men and women and over 70% of cases are preventable. A western diet, characterized by low vegetable and high red and processed meat intake, indisputably increases colon cancer risk. Heme, which gives red meat its color, is highly reactive, induces hyperproliferation and promotes DNA damage in the colon to a greater degree than any other red meat-associated carcinogen. Preclinical models indicate dietary chlorophyll, which gives green leafy vegetables their color, binds and stabilizes heme in the lumen, preventing genotoxicity. Additionally, data from our randomized controlled weight loss trial indicate increasing red meat consumption has deleterious effects on the gut microbiome, which is also implicated in colon cancer etiology. Because heme-containing foods are the richest sources of bioavailable iron and several other vitamins and minerals, mitigating their potential risks may be more beneficial than eliminating meat, poultry, fish and seafood in their entirety from the diet for risk reduction.

This feasibility study will begin to explore the research question: Will adding chlorophyll-rich green leafy vegetables to the diet prevent the deleterious effects of heme-rich red meat on the human host and microbiome? The investigators will randomly assign 50 adults at increased risk of colorectal adenoma to a block randomized crossover study with two 4-week dietary regimens in which: 1) participants will be provided with frozen green leafy vegetables and counseled to consume a high chlorophyll diet including 1 cup per day of cooked green leafy vegetables and normal meat (high heme) consumption; or 2) continue their normal high heme, low chlorophyll diet (control). A 4-week washout period encouraging habitual diet will be employed between the intervention periods and data will be collected at all four time points.

This study is critical in translating preclinical findings and has the potential to open the door to new knowledge and standards of care in colon cancer prevention. This study is a required step to aid in the design of a larger RCT to determine whether increased green leafy vegetable consumption mitigates the negative effects of red meat on DNA damage, inflammatory cytokines and gut microbe composition. This could lead to equally beneficial dietary guidance for colon health that might be more easily attained by the general public through addition, rather than omission of specific foods.

DETAILED DESCRIPTION:
Fifty thousand cases of colon and rectal cancer (CRC) could be prevented each year through screening, increased exercise and improved diet. Obesity alone increases risk of CRC by 33% and is associated with increased CRC mortality. Red and processed meat consumption is associated with increased CRC risk, most often in the context of dietary patterns, which juxtapose "Western" and "prudent" diets. A recent meta-analysis of 24 case control studies and 11 prospective cohort studies (n=1,295,063 men and women) found an 18% reduction in risk for colon cancer in the groups consuming the highest levels of cruciferous and green leafy vegetables. Risk reduction with high green leafy vegetable consumption remained significant regardless of whether pooled studies controlled for meat and/or total energy intake.

Heme-induced genotoxicity of the colon is prevented by chlorophyll in rodent models; an important finding that has not been tested in clinical trials though is supported by epidemiological observation.

This trial utilizes a crossover design to assess the feasibility of a dietary intervention in adults at increased risk of CRC. The overall intent of this line of research is to elucidate a CRC risk-reducing dietary pattern that is accessible to the general public. Therefore, obese, meat-eating participants will be randomized to an intervention and control diet: 1) high chlorophyll (green leafy vegetables) and high heme (normal meat) consumption; and 2) habitual high heme, low chlorophyll diet (control). During the intervention periods, all participants will receive individual dietary counseling from a registered dietitian two days per week to reinforce daily consumption goals based on the amounts of chlorophyll and heme in various foods. This study translates preclinical models, utilizes an appropriate at-risk population, and if feasible, has the potential to be tested for efficacy for the reduction of colon cancer risk.

Participants will be recruited through the Auburn University Pharmaceutical Care Clinic and throughout the Auburn community. After completing all baseline procedures, participants will be block randomized by gender due to potential differences in fecal microbiome. All participants will receive the intervention; the order in which it is received will be randomly generated. For the high chlorophyll study arm, a goal of 1 cup cooked dark leafy green vegetables will be prescribed, and participants will be instructed to consume at least ½ cup cooked dark green leafy vegetables during the same meal they consume red meat. The high chlorophyll group will also receive a variety of frozen dark green leafy vegetables, including, spinach, kale, collards, mustard greens, and turnip greens. Frozen vegetables are provided because flash-freezing minimizes nutrient loss and prevents chlorophyll degradation. Though the chlorophyll content varies between these species, it is exponentially higher than other green vegetables in the brassica family. Participants will be instructed to consume cooked vegetables, rather than raw, to increase the bioavailability of chlorophyll and reduce the volume of the needed amount of vegetable.

After each 4-week period, participants will complete questionnaires, return unused frozen vegetables (which will be tracked), provide a stool sample, and undergo phlebotomy. Study staff will obtain two 24-hour dietary recalls on non-consecutive days. Participants will be provided with an additional fecal collection kit for the sample that will be obtained prior to the next dietary arm assignment.

The behavioral framework of this intervention will utilize Social Cognitive Theory as the basis for behavior change in each intervention arm. Participants will increase self-efficacy of dietary adherence by setting goals and logging daily food intake (self-monitoring), which will be assessed in twice weekly counseling sessions with a registered dietitian.

ELIGIBILITY:
Inclusion Criteria:

* Consume less than 2 servings of green leafy vegetables per day
* Consume 5 or more servings of red meat per week
* BMI >30 kg/m2
* Agrees to not change dietary supplements during course of study
* Willing to comply with dietary regimen over course of study
* Able to store and cook frozen green leafy vegetables (freezer and microwave)
* Able to speak and read English

Exclusion Criteria:

* Previous diagnosis of colon cancer
* Use of any of the following in the past 4 weeks: systemic antibiotics, corticosteroids, immunosuppressive agents, commercial probiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Feasibility - accrual | 9 months
  Accrue 50 participants
Feasibility - retention | 12 weeks
  Retain 90% of sample at crossover and 80% at completion
Feasibility - adherence | 4 weeks during intervention phase
  Meet chlorophyll intake goals 90% of days

SECONDARY OUTCOMES:
DNA damage | Change from baseline to 4 weeks and 8 weeks to 12 weeks
  Serum 8-hydroxy-2'-deoxyguanosine
Inflammatory marker - C-Reactive Protein | Change from baseline to 4 weeks and 8 weeks to 12 weeks
  Serum hsCRP
Inflammatory marker - Tumor Necrosis Factor-alpha | Change from baseline to 4 weeks and 8 weeks to 12 weeks
  Serum TNF-alpha
Inflammatory marker - Interleukin 6 | Change from baseline to 4 weeks and 8 weeks to 12 weeks
  Serum IL-6
Gut microbe composition | Change from baseline to 4 weeks and 8 weeks to 12 weeks
  16s changes in microbiota alpha diversity
Bile acids | Change from baseline to 4 weeks and 8 weeks to 12 weeks
  Plasma primary and secondary bile acids
Body composition | Change from baseline to 4 weeks and 8 weeks to 12 weeks
  Body fat percentage using Bioelectrical Impedence Analysis
Acceptability | 4 weeks during intervention phase
  Acceptability of the diets will be measured by the Food Acceptability Questionnaire (FAQ) total score. The FAQ is a 10 item questionnaire scored on a 7-point likert scale with total scores ranging from 7-70.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Fruge, PhD, RD, Principal Investigator — Auburn University
Locations (1):
- Auburn University, Auburn, Alabama, United States

REFERENCES:
- [Background] Fruge AD, Ptacek T, Tsuruta Y, Morrow CD, Azrad M, Desmond RA, Hunter GR, Rais-Bahrami S, Demark-Wahnefried W. Dietary Changes Impact the Gut Microbe Composition in Overweight and Obese Men with Prostate Cancer Undergoing Radical Prostatectomy. J Acad Nutr Diet. 2018 Apr;118(4):714-723.e1. doi: 10.1016/j.jand.2016.10.017. Epub 2016 Dec 15. PMID 27988219
- [Background] Fruge AD, Van der Pol W, Rogers LQ, Morrow CD, Tsuruta Y, Demark-Wahnefried W. Fecal Akkermansia muciniphila Is Associated with Body Composition and Microbiota Diversity in Overweight and Obese Women with Breast Cancer Participating in a Presurgical Weight Loss Trial. J Acad Nutr Diet. 2020 Apr;120(4):650-659. doi: 10.1016/j.jand.2018.08.164. Epub 2018 Nov 9. PMID 30420171
- [Result] Fruge AD, Smith KS, Riviere AJ, Demark-Wahnefried W, Arthur AE, Murrah WM, Morrow CD, Arnold RD, Braxton-Lloyd K. Primary Outcomes of a Randomized Controlled Crossover Trial to Explore the Effects of a High Chlorophyll Dietary Intervention to Reduce Colon Cancer Risk in Adults: The Meat and Three Greens (M3G) Feasibility Trial. Nutrients. 2019 Oct 2;11(10):2349. doi: 10.3390/nu11102349. PMID 31581743
- [Derived] Riviere AJ, Smith KS, Schaberg MN, Greene MW, Fruge AD. Plasma and fecal zonulin are not altered by a high green leafy vegetable dietary intervention: secondary analysis of a randomized control crossover trial. BMC Gastroenterol. 2022 Apr 12;22(1):184. doi: 10.1186/s12876-022-02248-3. PMID 35413837
- See also: Meat and Three Greens website and link to eligibility survey — https://cws.auburn.edu/eatyourgreens/